CLINICAL TRIAL: NCT02475174
Title: Blood Circulation Assessment of the Superior Member in Women in Post-surgery for Breast Cancer Submitted to the Manual Lymphatic Drainage
Brief Title: Manual Lymphatic Drainage in the Superior Member in Women in Post-surgery for Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Elaine Caldeira de Oliveira Guirro, Lais Mara Siqueira das Neves, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HCRP nº 13408/2013
Record Dates: First submitted 2015-06-10; First posted 2015-06-18 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Without upper limb elevation (Experimental): Manual lymphatic drainage will be held with the voluntary supine without upper limb elevation.
  Interventions: Other: Without upper limb elevation
- Upper limb elevation to 30º (Experimental): Manual lymphatic drainage will be held with the voluntary supine with the upper limb elevation to 30º.
  Interventions: Other: Upper limb elevation to 30º

INTERVENTIONS:
Other: Without upper limb elevation — Lymphatic drainage without elevation of the upper limb.
  Arms: Without upper limb elevation
Other: Upper limb elevation to 30º — Lymphatic drainage with elevation of the upper limb to 30º.
  Arms: Upper limb elevation to 30º

SUMMARY:
Evaluate the effect of Manual Lymphatic Drainage (MLD) massage in arterial and venous circulation of the upper limb ipsilateral of women submitted after axillary lymphadenectomy breast cancer.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effect of Manual Lymphatic Drainage (MLD) massage in arterial and venous circulation of the upper limb ipsilateral of women submitted after axillary lymphadenectomy breast cancer. Will be evaluated 30 volunteers aged between 40 and 60 years, divided into 2 equal groups, submitted at MLD: Group 1 - volunteers who underwent surgery for breast cancer that have lymphedema, subject to manual lymphatic drainage without upper limb elevation; Group 2 - volunteers who underwent surgery for breast cancer that have lymphedema, subject to manual lymphatic drainage with the upper limb elevation to 30º. Data will be collected by ultrasound Doppler in vein and brachial artery before, after MLD, immediately after, and 30 minutes after therapeutic treatment, with and without elevation of 30°, cross over delimitation, being made a therapy session for therapeutic use with and without elevation, with interval period (washout) for seven days. The order of treatment protocols will be randomized by simple raffle for each volunteer. The data within and between groups will be evaluated by a statistical test t student or ANOVA. Otherwise it will be used Kruskal-Wallis followed test by Dunn. Data processing will be performed by software and fixed the critical level of 5% (p<0,05).

ELIGIBILITY:
Inclusion Criteria:

* Women with axillary lymphadenectomy surgery
* Lymphedema
* Aged 40-60 years.

Exclusion Criteria:

* Women with muscle-tendon injury and / or joint injuries member
* Skin disorders
* circulatory diseases.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-06 (Actual); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Blood flow velocity (Flow velocity in brachial artery and vein) | one day
  Flow velocity in brachial and artery vein

SECONDARY OUTCOMES:
Volume upper limbs | one day
  Volume upper limbs